CLINICAL TRIAL: NCT00850122
Title: An Open Label Study to Describe the Pharmacokinetics of Cefazolin in Preterm Neonates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phillip Brian Smith (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Phillip Brian Smith, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00012011; 1K23HD060040-01 (NIH)
Record Dates: First submitted 2009-01-22; First posted 2009-02-24 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Sepsis; Prematurity
MeSH Terms: conditions — Sepsis; Premature Birth | interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cefazolin (Experimental): Dosage Number of Infants
  ≤28 days of age 25 mg/kg IV q12 6 29-120 days of age 25 mg/kg IV q8 6
  Interventions: Drug: cefazolin

INTERVENTIONS:
Drug: cefazolin — Cefazolin dosing - administered for 48 hours Dosage
  ≤28 days of age 25 mg/kg IV q12 29-120 days of age 25 mg/kg IV q8

SUMMARY:
This is a phase I open label multi-dose study to investigative the pharmacokinetics and safety of cefazolin in infants <121 days of age and < 28 weeks gestation with suspected sepsis. There will be two cohorts of 6 infants each: 1) >48 hours of age and ≤28 days and 2) >28 days of age and <121 days of age. The study requires administration of the study drug over 2 days followed by 1 week of safety monitoring. Six 200 µL pK samples will be obtained over the 2 days of drug administration. The risks are reasonable vs. the benefits and have been minimized appropriately. There may be benefit to the subjects (administration of empirical antimicrobial therapy), and information from the study may benefit a large number of other infants in whom the drug is currently being administered despite the lack of PK data in this population.

ELIGIBILITY:
Inclusion Criteria:

* < 28 weeks gestation at birth
* > 48 hours and <121 days of age at the time of study drug administration
* One of the following:

  * Suspected systemic infection
  * Receiving cefazolin for prophylaxis
  * Receiving cefazolin treatment of a systemic infection

Exclusion Criteria:

* History of anaphylaxis attributed to a β-lactam
* Exposure to cefazolin in the month prior to study
* Serum creatinine > 1.7 mg/dL

Ages: 48 Hours to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2013-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Cefazolin pharmacokinetics including half life, clearance, and volume of distribution | Dose 1 and Dose 4

SECONDARY OUTCOMES:
Safety | 7 days following last dose of cefazolin

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, Brazil